CLINICAL TRIAL: NCT04570566
Title: Evaluation of Horizontal Alveolar Ridge Augmentation Using Pericardial Membrane Versus Titanium Mesh" Histological and Clinical Study
Brief Title: Comparison Using Pericardial Membrane Versus Titanium Mesh" in Horizontal Alveolar Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Wafaa Abaza, general practitioner, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-REC IM021726
Record Dates: First submitted 2020-09-21; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Horizontal Ridge Augmentation, Histological and Clinical Result

STUDY DESIGN:
Intervention Model Description: The present randomized clinical study was conducted to assess histological, histomorphometric, radiographic and the clinical response of bone after 4 months of augmentation and to compare the amount of horizontal bone gained between both groups and compare the quality of gained bone using a native pericardium physical resorbable barrier made of bovine pericardium with 1:1 mixture of bone graft in test group versus using titanium mesh with 1:1 mixture of bone graft in control group to augment localized horizontal alveolar ridge defects for the subsequent placement of dental implants.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- titanium mish (Experimental): horizontal alveolar ridge augmentation with non-resorbable titanium mish .evaluation after 4 months
  Interventions: Procedure: horizontal alveolar ridge augmentation
- pericardium membrane (Experimental): horizontal alveolar ridge augmentation with resorbable pericardium membrane then .evaluation after 4 month.
  Interventions: Procedure: horizontal alveolar ridge augmentation

INTERVENTIONS:
Procedure: horizontal alveolar ridge augmentation — evaluate the potential application of resorbable pericardium membrane to augment localized alveolar ridge defects in esthetic zone, from histological, radiographical and clinical aspects in comparison with titanium mish for the subsequent placement of dental implants

SUMMARY:
Randomized clinical trial study ,The purpose of this study To evaluate the potential application of resorbable pericardium to augment localized alveolar ridge defects in esthetic zone, from histological, radiographical and clinical aspects in comparison with titanium mish for the subsequent placement of dental implants Reconstruction of alveolar bone defect can be achieved through many regenerative surgical procedures including guided bone regeneration (GBR).Tenting of the periosteum using a cortical bone block maintains space and minimizes resorption of the particulate graft volume

DETAILED DESCRIPTION:
Randomized clinical trial study ,The purpose of this study To evaluate the potential application of resorbable pericardium to augment localized alveolar ridge defects in esthetic zone, from histological, radiographical and clinical aspects in comparison with titanium mish for the subsequent placement of dental implants Reconstruction of alveolar bone defect can be achieved through many regenerative surgical .

Patient selection:

20 patients will be selected from the outpatient clinic of the department of, Oral medicine and Periodontology, Faculty of Dentistry, Ain Shams University.

Patient grouping and treatment protocol The purpose of this study is to evaluate the results of alveolar ridge augmentation using two types of guided membranes.

Patients will be randomly divided into two groups according to the type of membrane will used in alveolar ridge augmentation.

All the patient's records will be coded, known only by the researcher for the purpose of confidentiality.

Every patient participating in this study will sign an informed consent demonstrating the purpose of this study, surgical procedure, probable risks and benefits from this surgical intervention.

In case of failure, the patient will be compensated with the suitable ordinary either fixed or removable prosthesis. Every patient could quit at anytime without penalty or loss of any benefits. The faculty research ethics committee will review the proposal.

Eligible patients will be randomized in a 1:1 ratio into two groups; (Group I) included 10 patients and (Group II) included 10 patients. The computer-generated randomization assignment (blocks of 4) and allocation concealment will be performed by sealed envelopes containing the randomization number prepared by non involved member and sent to principle investigator to assign the interventions to patients.

Group 1:

Will include 10 patients and alveolar ridge augmentation will be performed using intraoral autogenous block bone graft in addition to particulate xenograft to fill discrepancies covered by titanium mesh .

Group 2 Will include 10 patients and alveolar ridge augmentation will be performed using intraoral autogenous block bone grafting addition to particulate xenograft to fill discrepancies covered by pericardial membrane.

Patients may suffer postoperatively from pain, edema, infection which will be controlled by antibiotics and anti-inflammatory and proper oral hygiene measures with chlorhexidine mouth wash.

Risks of failure will be minimized as much as possible by proper patient selection, properly prepared surgical protocol, and rapid placement of the graft after harvesting to avoid viable cells death, short surgeries as much as possible, strict aseptic techniques, proper infection control measures, proper home oral hygiene measures and regular follow ups for maintenance of the oral hygiene.

Measurements and evaluation of edentulous ridge

* Preoperative evaluation will be performed for all patients at baseline. This evaluation will include Cone Beam Computed Tomography (CBCT) using standardized and clinical photographs using UNC periodontal probe .
* Two different techniques will be used to measure the alveolar ridge labiolingual width before and after ridge augmentation:

  1. Cone Beam Computed Tomography (CBCT)

This will be carried out at 2 intervals:

1. Baseline CBCT will be performed before the first surgery.
2. The second CBCT will be performed before the second surgery.

The Ridge measurement technique will standardized by using vacuum form acetate stent (0.4 mm base plate thermoforming material). references points placed on palatine surface using gutta-percha point .t this point sagittal section of the ridge has taken on CBCT software ,same stent used during 2nd cone beam after 4 months and take a sagittal section cut at level of same gutta percha point : at same sagittal cut which taken at pre and post operative cone beam measuring a horizontal Bucco -lingual line width on 3 points occlusal-apical .

2-UNC 15-color coded probe

1. at first surgery; done on the bony ridge directly after mucoperiosteal flap elevation before bone graft placement.
2. During the second surgery (re-entry surgery for implant placement) after 4 months; it will be done on the bony ridge with the mucoperiosteal flap elevation.

   .

   Evaluation of the Augmented Bone Quality:

   After 4 month re-entry for implant placement and histological evaluation of the grafted bone should be performed.

   Preoperative preparation:

   The surgical procedures were performed under local anesthesia of Articainchlorhydrate1:100000.

   Pre-operative rinsing of the oral cavity with a 0.2% chlorhexidine and a perioral skin disinfection with Betadine antiseptic solution. An antibiotic therapy 1 h before surgery will administrated to the patient, with 2 g of amoxicillin clavulanate (Augmentin)

   Incision and preparation of recipient site:

   A mid-crestal horizontal incision will be made with oblique releasing incisions where needed in order to mobilize a full-thickness flap.

   The flap will carefully be elevated from the palatal and buccal aspect of the alveolar ridge.

   All the granulation tissue will be removed from the cortical bone. The intra-surgical evaluation confirmed a narrow alveolar ridge with insufficient crest width for ideal dental implant placement gauged by using UNC 15-color coded periodontal probe or bone caliber caliper to identify and measure the greatest horizontal alveolar ridge defect.

   Intra-surgical evaluation confirmed a narrow alveolar ridge with insufficient crest width for ideal dental implant placement

   Perforations into the marrow space will performed using small round surgical burs to facilitate vascularization of the graft and cell colonization from the bone marrow.

   Bone graft From Donor site:

   For both groups:
   * Sub-marginal attached gingival incision will be used for papilla preservation
   * The intraoral autogenous block graft will be harvested from the mandible symphyses using trephine burs.
   * The donor site will be examined clinically and radiographically, it should be easily accessible, with no apparent infection or anatomical abnormality .

   In cases Guided Bone Regeneration with Titanium mesh ( Ti-mesh):
   * A 0.2 mm thickness Ti-mesh will be trimmed and adapted to the surgical defect to create a proper bone contour.
   * The Ti-mesh should be shaped avoiding sharp edges in order to prevent soft tissue dehiscence or exposure.
   * The minimum distance from the periodontium of the neighboring teeth was 1.5 mm in order to prevent possible infiltrations through the gingival sulcus
   * The defects will be filled with autogenous bone block, bone chips mixed with xenograft , so that the deficiencies completely filled, this will recreate the ideal amount of bone for subsequent implant placement.
   * The Ti-mesh then placed over the graft and fixed to the palatal and buccal bony walls using cortical screws on each side to prevent any micro movement.
   * Periosteal incisions on the flaps will be performed in order to promote a tension-free closure and to mobilize the buccal flap and obtain the passive closure essential to prevent dehiscence and Ti-mesh exposure.The releasing incisions should be placed 3 to 4 mm in length at the apical extent of the vertical releasing incision (in the buccal vestibule), which directed away from the vertical incisions created a split-thickness flap past the mucogingival line as they proceeded apically to release the flap
   * Double layer suture should be applied with horizontal mattress and circumferential interrupted suture using a suture 5-0 polypropylene suture, to seal the overlapping periosteal portion of the palatal and buccal flap.

   In cases of Guided Bone Regeneration using pericardium membrane with tenting screw:
   * The augmentation technique will used in both treatment groups is the same, with the exception of the membrane material.
   * 1.4-mm-diameter titanium reference screw will be placed perpendicular to the alveolar ridge, extending laterally to the desired amount of horizontal augmentation and fixed the autologous bone block which act as tenting with titanium screw.
   * The attempted horizontal gain will be measured, from the screw head to the bone using a UNC-15 periodontal probe.

   The particulate graft consisted of a combination of xenograft and particulate autogenous bone then applied to the recipient site using a bilayer technique with the autogenous particles placed against the native bone.
   * The particulate bone graft will be placed around supporting tenting screws to the level of the screw heads and covered with a pericardium membrane, which will be fixed to the bone with titanium tacks.
   * Primary closure should be obtained by using a combination of interrupted and horizontal mattress sutures using 5-0 polypropylene sutures, to seal the overlapping periosteal portion of the palatal and buccal flaps.

   Post-operative Medication and follow up:
   * 1 g of Augmentin twice a day for 7 days, 500mg metronidazole twice a day for 7 days, a 0.2% Chlorhexidine gluconate (mouthwash rinse solution 1min three times a day for the same period of time, starting the day after the surgery and Brufen 600 mg 3 times daily for 7 days as analgesic and anti inflammatory
   * The sutures will be removed after 14 days.
   * Follow up phase: 7 days after 1st surgery, fourteen days after the sutures will be removed then the patient will be instructed to return for follow-up visits every 2 weeks for the first month then once monthly until re-entry surgery. At the follow up visits both recipient and donor sites will be clinically examined for soft tissue healing .
   * After 4 months The second radiographic evaluation of alveolar ridge width by Cone Beam Computed Tomography (CBCT) will be performed before the second surgery.

     2nd surgical stage
   * Fixation and tenting screws which had been used to stabilize the graft during healing will be removed and retrieve the Titanium mesh.
   * A bone biopsy will be harvesting from the grafted area using trephine bur will obtained prior to implant placement for histological evaluation.
   * Implant placement.
   * All the patients will receive supra-structure prosthetic part .

   Statistical Analysis:

   All the clinical, Radiographical , Histomorphometric data will be tabulated and the result will be subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

Adult patients of both sexes. Healthy adult patients; all patients were free from any systemic diseases as evidenced Burkitt's Oral Medicine health history questionnaire Age from 20-50 years old. partially edentulous area in upper arch esthetic zone (incisors to premolar area). Residual bone width ≤4 mm and minimum alveolar vertical dimension measured ≥8 mm from the alveolar crest to the roof of the nasal cavity or maxillary sinus, (H.2.e) (Cologne Classification 2013).

Exclusion Criteria:

Subjects with any systemic disease or conditions according to health questionnaire assessment modified from oral medicine .

uncontrolledly diabetic HBAc1 more than 8 history of base phosphonate medication history of radiotherapy medication Active periodontal disease. Smokers more than 5 cigarettes per day Pregnant and breastfeeding females . Mentally retarded patients. Vulnerable groups (prisoners, mentally disabled, and decision impaired individuals).

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Histological | 4 months
  histomorphometric evaluation of the grafted boneThe area fraction (AF) of newly formed bone was measured automatically. The area fraction represents the percentage of the newly formed bone trabeculae to the total area of the microscopic field. The mean area fraction (MAF) for each case was calculated. Estimation of osteocytes count in each microscopic field, viable osteocytes within their lacunae in the newly formed bone

SECONDARY OUTCOMES:
clinical | 4 months
  Radiographic evaluation of alveolar ridge bucco-lingually dimensional changes following alveolar ridge augmentation using Cone Beam Computed Tomography.
clinical | 4 months
  Clinical evaluation of alveolar ridge dimensional changes following alveolar ridge augmentation using UNC-15 mm periodontal prob

CONTACTS AND LOCATIONS:
Overall Officials: Nevine A Hassan Kheir El Din, professor, Study Director — Ain Shams University
Locations (1):
- faculty of dentistry Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided